CLINICAL TRIAL: NCT03740295
Title: Impact of Ketone Bodies and Epigallocatechin Gallate in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Collaborators: Valencian Institute of Neurorehabilitation Foundation (Unknown)
Responsible Party: Principal Investigator, José Enrique de la Rubia Ortí, Director, Fundación Universidad Católica de Valencia San Vicente Mártir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FundacionUCV
Record Dates: First submitted 2018-10-05; First posted 2018-11-14 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Coconut Oil; epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Multiple Sclerosis (Placebo Comparator)
  Interventions: Other: Placebo
- Intervention Multiple Sclerosis (Experimental)
  Interventions: Dietary Supplement: Coconut oil and epigallocatechin gallate

INTERVENTIONS:
Dietary Supplement: Coconut oil and epigallocatechin gallate — 600 mg of epigallocatechin gallate (EGCG) and 60 ml of coconut oil (3600 mg of TGCM) per day, divided into two doses (one in the morning and one at noon)
  Arms: Intervention Multiple Sclerosis
Other: Placebo — Lactose
  Arms: Control Multiple Sclerosis

SUMMARY:
Based on the fact that the fundamental pathogenic mechanism of the Multiple Sclerosis (MS) disease is neuroinflammation, related in turn to cellular oxidation and mitochondrial alterations, this project aims to assess the impact of a nutritional intervention on the evolution of MS patients in their different slopes. To this end, the administration of medium-chain triglycerides, whose metabolism produces the increase of ketone bodies in the blood, will be carried out; and another of the antioxidant polyphenol epigallocatechin gallate. This procedure will be applied over 6 months, based on a isocaloric Mediterranean diet, with a population for the study of 80 patients with different variants of the disease. The assessment of the intervention will be carried out every two months, at motor-functional, anthropometric, cognitive and emotional, inflammatory, and oxidation levels.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis patients older than 19 years ans under 65 who sign informed consent of the study

Exclusion Criteria:

* Patients with coconut oil intolerance or other chronic metabolic pathologies

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Lipid peroxidation Malondialdehyde (MDA) | 0-4 months
  Malondialdehyde (MDA) will be used as perioxidation marker. It is based on the reaction of thiobarbituric with malondialdehyde, product of the splitting of hydroperoxides, thus forming a color that can be measured directly. Its analysis is used for its good practicability and simplicity, but it lacks sensitivity, so it is recommended, to increase it, to use fluorometric or chromatographic procedures.
Tumor necrosis factor alfa (TNF-alpha) | 0-4 months
  Plasma concentrations of inflammatory markers (IL-6 and TNF-a) were determined by using a multiplex ELISA (Human ProInflammatory II 4-Plex Ultra-Sensitive Kit; Meso Scale Diagnostics).
Interleukin 6 (IL-6) | 0-4 months
  Plasma concentrations of inflammatory markers (IL-6 and TNF-a) were determined by using a multiplex ELISA (Human ProInflammatory II 4-Plex Ultra-Sensitive Kit; Meso Scale Diagnostics).

SECONDARY OUTCOMES:
Quantitative electroencephalogram (QEEG) | 0-4 months
  A QEEG brain map (or 'Q' for short) enables us to see your unique pattern of mental strengths and weaknesses - areas of the brain where there is too little or too much activity, and areas that are not coordinating their activity the best they could.
Betahydroxybutyrate | 0-4 months
  Beta-hydroxybutyrate (BHB) inhibits the NLRP3 gene, which is part of a complex set of proteins called the inflammasome.
  The inflammasome drives the inflammatory response in several diseases, among which are some autoimmune diseases.
C-reactive protein | 0-4 months
  C-reactive protein (CRP) is produced by the liver. The level of CRP rises when there is inflammation throughout the body. This is one of a group of proteins called "acute phase reactants" that increase in response to inflammation.
Haptoglobin | 0-4 months
  Haptoglobin is an acute phase protein whose expression is a response proportional to inflammation
Field oxide (FOX) | 0-4 months
  The method is based on the principle of the rapid peroxide-mediated oxidation of Fe2+ to Fe3+ under acidic conditions.
Total antioxidants (TEAC) | 0-4 months
  TEAC is a spectrophotometric technique that is based on inhibition from the antioxidants of the absorbance of the radical cation of 2,2'-Azino-bis(3-ethylbenzothiazoline-6-sulfonic acid) diammonium salt (ABTS) (2,2'-azinobis (3-ethylbenzothiazoline-6-sulfonate), a stable blue-green chromophore that has a characteristic long wavelength absorption spectrum
Copper reduction capacity (CUPRAC) | 0-4 months
  CUPRAC method based on the reduction of Cu (II) in hydroetanolic medium (pH 7.0) in the presence of neocuproin (2,9-dimethyl-1,10-phenanthroline), by polyphenols resulting in complexes of Cu.
Iron reduction capacity (FRAP) | 0-4 months
  The FRAP assay, is presented as a novel method for assessing ''antioxidant power.'' Ferric to ferrous ion reduction at low pH causes a colored ferrous-tripyridyltriazine complex to form.
Paraoxonase 1 (PON1) | 0-4 months
  The enzyme Paraoxonase 1 (PON-1), is synthesized in the liver and is attached to the apolipoprotein A1 of high density lipoprotein (HDL). PON1 is able to hydrolyze organophosphates compounds (e.g. paraoxon, diazoxon, soman, sarin), has arylesterase and lactonase function by hydrolyzing lactones, homocysteine thiolactone specifically to regenerate homocysteine.
Anxiety | 0-4 months
  The State-Trait Anxiety Inventory (STAI). This is a self-report measure of immediate and general anxiety. A patient is shown or read aloud a statement (e.g. 'I feel jittery') and is required to indicate to what degree, from a choice of four frequencies, the statement relates to them. Range score for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the State Anxiety.
Depression | 0-4 months
  Beck Depression Inventory (BDI). This is a self-report measure of depression. A patient is shown or read aloud groups of four statements, which range from a normal thought to a profoundly depressed thought. The patient must indicate which of the four is closest to how they have been feeling over the past week. The range score is 0-63, the higher score indicating greater depression.
Satiety | 0-4 months
  Perceptions of hunger, desire to eat and satiation were performed by VAS, which provides an accurate way to predict appetite in young adults and has good reproducibility. VAS, 100mm in lenght with words anchored at each end, expressing the most positive and the most negative rating, were used to assess hunger, satiety, fullness, prospective food consumptions best represented their sensation at the time. The volunteers were instructed to make a point at the point where best represented their sensation at the time.
Sociodemographic | 0 months
  The demographic characteristics (age, gender, etc.) and clinical characteristics (year of diagnosis, type of multiple sclerosis, etc.) of the sample were measured through an ad hoc sociodemographic questionnaire.
Berg | 0-4 months
  This scale rates performance from 0 (cannot perform) to 4 (normal performance) on 14 items with a maximum total score of 56.18,19 The validity and reliability of the scale have been assessed on populations of subjects with multiple sclerosis.
Exercise tolerance | 0-4 months
  The Two-minute walk test (2MWT) is a short version of an exercise tolerance test and reports the distance in meters during a 2-minute walk. The objective of the test is to walk as far as possible for 2 minutes. Participants, remembering the objective, walked at a comfortable speed between 2 cones that were 20m apart. If they had to turn, they moved the unaffected side. They were permitted to slow down, stop, and rest as necessary during the 2-minute walk. The time was started when participants started walking and proceeded until 2 minutes elapsed, even if they slowed down or stopped walking. The instructions were, "Go. Keep walking until I say 'stop' or until you are too tired, and stop when I say 'stop.'"
Gait speed | 0-4 months
  The 10-meter walk test is a simple, effective and widely used tool to evaluate gait speed. The 6MWT evaluates endurance by measuring the maximum distance an individual can walk within 6 min, and determines the walking capacity.
Physical function and symptoms | 0-4 months
  Disabilities of the arm, shoulder and hand (DASH) 30 items, self-report rating scale will be used to measure physical functions and symptoms' in people with disorders of the upper limb. Items are scored from 1 (no difficulty) to 5 (unable). A total 'disability/symptom' score is generated by summing items, and averaging to produce a mean item score between 1 and 5. This value is then transformed to a score out of 100 by subtracting one and multiplying by 25. A higher score indicates greater disability.
Neurological impairment | 0-4 months
  Kurtzke's Expanded Disability Status Scale (EDSS) is the most widely used measure which attempts to capture the full extent of MS symptoms in a standardised way. It was selected for this study because of its universal currency. Both the EDSS and Functional Systems were recorded. The EDSS provides a total score on scale that ramges from 0 to 10. The higher degrees means more disability.
Manual dexterity | 0-4 months
  It was measured with the Nine Hole Peg Test (NHPT). The time needed to place and remove 9 pegs was recorded and averaged over 2 trials. Manual dexterity speed was calculated as pegs per second and used in the analyses. Participants who were not able to place any peg within a time limit of 300 seconds received a score of 0 pegs per second.
Hand Grip Strength | 0-4 months
  The instrument used was a Jamar handgrip dynamometer. The dynamometer has a dial meter. Its handle was positioned in the second notch. In that position the grip width was approximately 4.0 cm
Muscle power | 0-4 months
  The muscle scale qualifies muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle.
Muscle Strength Assessment Dynamometer (NEDDFM/IBV ) | 0-4 months
  This allows the determination of the degree of muscular weakness of the large muscular groups of lower and upper limb in the different planes of movement.
  The system assists the evaluator, providing, in real time, the force exerted by a certain muscle group, the maximum effort reached during the exercise and the corresponding deficiency according to the scales of RD 1971/1999 or the AMA disability assessment tables. The results of the assessment can be displayed on the screen and printed on a report card.
Body diameters | 0-4 months
  Distance taken in projection, between two anatomical points and measured in centimeters (cm), through a pachymeter.
Body perimeters | 0-4 months
  They are indicators of body fat and protein reserves, so they are useful to know the nutritional status. Perimeters from the thorax, waist, arm, forearm and thigh, will be measure in centimeters (cm), through a tape measure.
Skinfold calipe | 0-4 months
  This method is based on the measurement of the thickness of the subcutaneous adipose tissue in precisely defined and protocolized places, measured with a pleximeter and taking into account the guidelines of the ISAK (The International Society for Advancement of Kinanthropometry).
Height | 0-4 months
  It is expressed in centimeters (cm), measuring the distance between the vertex and the plane of support of the individual by means of a stadiometer and placing the head on the Frankfort plane
Weight | 0-4 months
  Sum of fat mass and lean mass, expressed in kilograms (kg) and measured by clinical scale.

CONTACTS AND LOCATIONS:
Locations (1):
- José Enrique de la Rubia Ortí, Valencia, Spain